CLINICAL TRIAL: NCT07246109
Title: The Effects of Knee Brace and Muscle Training on Osteoarthritis Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Screening
Other Study IDs: CMUH-113-REC3-182; china medical university (Other: china medical university and hospital)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis (OA) of the Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New brace (Experimental): wearing a new knee brace for 4weeks
  Interventions: Device: knee brace
- Traditional knee brace (Sham Comparator): wearing a traditional knee brace for 4weeks
  Interventions: Device: knee brace

INTERVENTIONS:
Device: knee brace — This research will employ a randomized single-blind crossover trial to compare the effectiveness of the new and traditional braces. This project will utilize various evaluation tools, including pain scales, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), participant satisfaction, muscle tension, Q-angle measurements, and joint range of motion. This project will assess the impacts of the new knee brace and BFR in alleviating pain and improving mobility.

SUMMARY:
A new non-weight-bearing knee brace has been developed to correct abnormal alignment and reduce joint pressure, showing promising results in alleviating knee osteoarthritis symptoms compared to traditional braces. In addition, Blood Flow Restriction (BFR) training, which involves using pressure bands to simulate high-intensity exercise during low-intensity workouts, has been shown to enhance muscle strength.

This research will employ a randomized single-blind crossover trial to compare the effectiveness of the new and traditional braces, while also assessing BFR's impact on lower limb strength and knee function. This project will utilize various evaluation tools, including pain scales, Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), participant satisfaction, muscle tension, Q-angle measurements, and joint range of motion. This project will assess the impacts of the new knee brace and BFR in alleviating pain and improving mobility.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers over 50 years of age who are able to fully comply with the study procedures.

Subjects diagnosed with unilateral or bilateral knee osteoarthritis by a physician based on X-ray findings and clinical symptoms.

Radiographic diagnosis is evaluated using the Kellgren and Lawrence Scale (K/L grade) as the radiographic assessment tool.

Clinical diagnosis follows the American College of Rheumatology (ACR, 1991) criteria, which include clinical symptoms in combination with radiographic or laboratory findings.

The diagnostic criteria are:

1. Knee pain on most days of the past month.
2. Presence of osteophytes on X-ray.
3. Synovial fluid that is clear, viscous, and contains fewer than 2,000 white blood cells/mL.
4. Age over 50 years.
5. Morning stiffness of the knee lasting less than 30 minutes.
6. Crepitus on knee motion.

Diagnosis of knee osteoarthritis is confirmed when any of the following combinations are present:

Exclusion Criteria:

* Individuals with general contraindications to treatment, such as severe medical conditions, recent major trauma, or pregnancy.

Individuals with a history of substance abuse (including excessive alcohol consumption) that could affect pain perception.

Individuals with local skin infections, ulcers, or lesions in the treatment area.

Individuals who have undergone previous knee surgery or total knee arthroplasty.

Individuals with central or peripheral nervous system disorders.

Individuals with cognitive impairment who are unable to comply with the study procedures.

Individuals currently receiving other treatments for knee osteoarthritis.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index | up to 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan